CLINICAL TRIAL: NCT00699270
Title: A Prospective, Non-Controlled, Clinical Investigation of the Comprehensive®, BioModular®, and Bi-Angular® Shoulder Systems
Brief Title: A Clinical Investigation of the Comprehensive®, BioModular®, and Bi-Angular® Shoulder Systems
Status: Withdrawn | Type: Observational
Why Stopped: Business need changed.
Sponsor: Biomet Orthopedics, LLC (Industry)
Responsible Party: Sponsor
Organization: Zimmer Biomet (Industry)
Other Study IDs: Biomet 12380-76
Record Dates: First submitted 2008-06-13; First posted 2008-06-17 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Osteoarthritis; Avascular Necrosis; Rheumatoid Arthritis; Humeral Fractures
Keywords: Total Shoulder Arthroplasty; Total Shoulder Replacement; Shoulder Arthritis
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Arthritis, Rheumatoid; Humeral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomet Humeral Stems: Biomet Humeral Stems: Comprehensive®, BioModular®, and Bi-Angular® Shoulder Systems

SUMMARY:
The purpose of this prospective clinical data collection is to document the performance and clinical outcomes of Biomet Humeral Stems

ELIGIBILITY:
Inclusion Criteria:

* Non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis
* Rheumatoid Arthritis
* Correction of functional deformity

Exclusion Criteria:

Absolute contraindications:

- Infection, Sepsis, and Osteomyelitis

Relative contraindications:

* Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions
* Osteoporosis
* Metabolic disorders which may impair bone function
* Osteomalacia
* Distant foci of infections which may spread to the implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have already made the decision to undergo shoulder replacement surgery and will receive a Biomet humeral stem.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
UCLA End Result Score | 3 months, 6 months, 1 year, 3 years, 5 years
X-rays | 3 month, 1 year, 3 years, 5 years

SECONDARY OUTCOMES:
Incidence of revisions and removals | Any time

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth J Beres, MD, Study Director — Clinical Research, Biomet Orthopedics, LLC